CLINICAL TRIAL: NCT01823315
Title: A Multicenter, Prospective, Randomized Trial of Methotrexate Single-dose Treatment and Methotrexate/Actinomycin-D Single-dose Treatment in Low-Risk Gestational Trophoblastic Neoplasia
Brief Title: Methotrexate Single-dose Treatment and Methotrexate/Actinomycin-D Single-dose Treatment in Low-Risk Gestational Trophoblastic Neoplasia
Acronym: GTN-01
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ding Ma (Other)
Collaborators: Zhejiang University (Other); Huazhong University of Science and Technology (Other); Shandong University (Other)
Responsible Party: Sponsor-Investigator, Ding Ma, Director of the department of Obstetrics and Gynecology, Tongji Hospital, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-GYN/GTN-01
Record Dates: First submitted 2013-03-21; First posted 2013-04-04 (Estimated); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Gestational Trophoblastic Disease; Gestational Trophoblastic Neoplasia; Gestational Trophoblastic Tumor; Gestational Trophoblastic Neoplasms
MeSH Terms: conditions — Gestational Trophoblastic Disease | interventions — Dactinomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Methotrexate Single-coure chemotherapy (Experimental): Regimen: Methotrexate 0.4mg/(kg·d) intramuscularly (IM) on days 1-5. If 10-fold fall of hCG achieved 18 days after treatment completion, success of primary single-course chemotherapy was defined and further treatment was withheld; otherwise, failure was defined and the patient was referred to multi-course chemotherapy. During the period of observation for those with success, if the level of hCG became stationary for at least 3 weeks or rose again, the patient was also referred to multi-course chemotherapy. Additional consolidation chemotherapy with 1-3 courses was given for those who achieved CR by multi-course chemotherapy, but not by single-course regimen.
  Interventions: Drug: MTX 1
- Methotrexate+dactinomycin Single-dose chemotherapy (Experimental): Regimen: dactinomycin d 0.6mg/m2, IV, on day1, 2; methotrexate 100mg/m2, IV, on day1 (after Act-d); methotrexate 200mg/m2, IVgtt, on day1 (after methotrexate, 500ml NS, >4h).
  If 10-fold fall of hCG achieved 18 days after treatment completion, success of primary single-course chemotherapy was defined and further treatment was withheld; otherwise, failure was defined and the patient was referred to multi-course chemotherapy. During the period of observation for those with success, if the level of hCG became stationary for at least 3 weeks or rose again, the patient was also referred to multi-course chemotherapy. Additional consolidation chemotherapy with 1-3 courses was given for those who achieved CR by multi-course chemotherapy, but not by single-course regimen.
  Interventions: Drug: MTX 2; Biological: Act-d
- MTX multiple courses chemotherapy (Active Comparator): Regimen: methotrexate 0.4mg/(kg·d) intramuscularly (IM) on days 1-5, 2-week intervals. Patients continue on treatment until 1 beta HCG titer is below the institutional normal. Patients then receive at least 1 additional consolidation treatment.
  After treatment, all the patients were asked for contraception with condom or oral contraception. Regular hCG surveillance, once a month for 3 consecutive months and once every 3 months for 2 years, was performed. During follow-up period, pelvic ultrasound and pulmonary X ray or CT scan were conducted if needed.
  Interventions: Drug: MTX 1

INTERVENTIONS:
Drug: MTX 1 — MTX 0.4mg/(kg·d) intramuscularly (IM) on days 1-5
  Arms: MTX multiple courses chemotherapy; Methotrexate Single-coure chemotherapy
Drug: MTX 2 — MTX 100mg/m(2), IV, on day1 (after Act-d); MTX 200mg/m(2), IVgtt, on day1 (after MTX, 500ml NS, >4h)
  Arms: Methotrexate+dactinomycin Single-dose chemotherapy
Biological: Act-d — Act-d 0.6mg/m(2), IV, on day1,2
  Arms: Methotrexate+dactinomycin Single-dose chemotherapy

SUMMARY:
The investigators conducted a trial to determine whether methotrexate or methotrexate/dactinomycin single-course treatment work well as multiple courses of single methotrexate chemotherapy in low-risk gestational trophoblastic neoplasia. It is not yet known whether single-course of chemotherapy is as the same effectiveness as multicourse.

ELIGIBILITY:
Inclusion Criteria:

* Patients who FIGO Stage I, II, or III criteria for low-risk gestational trophoblastic neoplasia (GTN);
* WHO risk score 0-6;
* Age≤60 years; female, Chinese women;
* Initial treatment is chemotherapy; patients who received prior low-dose methotrexate for treatment of an ectopic pregnancy will be eligible for this study;
* Performance status: Karnofsky score≥60;
* Laboratory tests: WBC≥3.5×10(9)/L, ANC≥1.5×10(9)/L, PLT≥80×10(9)/L, serum bilirubin≤ 1.5 times the upper limit of normal, transaminase≤ 1.5 times the upper limit of normal, BUN, Cr≤ normal
* Provide written informed consent.

Exclusion Criteria:

* Patients with unconfirmed diagnosis of GTN;
* Patients with placental-site trophoblastic tumor (PSTT) or epithelioid trophoblastic tumor (ETT)
* WHO risk score >6;
* With severe or uncontrolled internal disease, unable to receive chemotherapy;
* Concurrently participating in other clinical trials
* Unable or unwilling to sign informed consents;
* Unable or unwilling to abide by protocol.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2012-12; Primary Completion 2015-12 (Actual); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) by single-course | through study completion, an average of 1 year
Completely remission rate by multiple courses after single-course failure | through study completion, an average of 1 year

SECONDARY OUTCOMES:
remission rate of ACTD replacement after MTX resistance | through study completion, an average of 1 year
the number of courses needed to achieve complete remission after multi-course treatment | through study completion, an average of 1 year
complete remission rate by multidrug combination therapy after single drug failure | through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Xing Xie, MD, PhD, Study Chair — Zhejiang University
Locations (3):
- China (3):
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Qilu Hospital，Shandong University, Jinan, Shandong
  - Women's Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang